CLINICAL TRIAL: NCT01628822
Title: Pilot Study, Prospective, Single Center,Randomized, Single Blind, Evaluating the Efficacy of Relaxation to 12 Weeks Against Placebo, in the Overall Care Chronic Pain in Patients With Fibromyalgia
Brief Title: Efficacy Study of Relaxation to 12 Weeks Against Placebo in the Overall Care Chronic Pain in Patients With Fibromyalgia
Acronym: Sophrodol-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOL11-DR-SERRA; 2011-A01055-36 (Other: ID-RCB)
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Relaxation; Improving the quality of life
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active relaxation (Experimental)
  Interventions: Behavioral: Active relaxation
- Placebo relaxation (Placebo Comparator)
  Interventions: Behavioral: Placebo

INTERVENTIONS:
Behavioral: Active relaxation — The length of follow-up will be 12 weeks.Patients will be seen once every seven days by a relaxation therapist for 5 weeks (6 sessions) and will be followed by the center physician investigator regarding drug therapy
  Arms: Active relaxation
Behavioral: Placebo — Patients are been asked to relax alone in a quiet room. They are coming every 7 days for 5 weeks (6 sessions) and will be followed by the investigator regarding drug therapy
  Arms: Placebo relaxation

SUMMARY:
The main objective of this protocol is to measure the improvement of the overall situation of patients with diffuse chronic pain or fibromyalgia to 12 weeks by non-drug treatment relaxation.

Secondarily,is to evaluate the evolution of physical variables, psychological and social improvement of the quality of life. To evaluate the evolution of drug consumption

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years
* established diagnosis of fibromyalgia as defined by the American College of Rheumatology: widespread pain and eleven tender points at 18 sites listed (ACR, 1990)
* EVA ≥ 4 (on a scale of 10 cm)
* no change in treatment for 15 days, except for treatment "on demand" or "rescue"
* patient has given its written consent
* patient wishing to benefit from relaxation sessions
* people who can meet the self-assessment and hetero-assessment
* people with a social security number

Exclusion Criteria:

* any painful situation that cannot be distinguished from fibromyalgia pain by the patient
* patients untreated or treated for less than a month
* patient with psychosis or severe depression or severe anxiety or impulsivity characterized, at the discretion of the clinician.
* patients receiving benzodiazepines at the request
* patient with deafness
* patient after a body treatment using a relaxation method, relaxation therapy or hypnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
scores on Fibromyalgia Impact Questionnaire (FIQ) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SERRA Eric, Dr, Principal Investigator — Activity Centre "Pain", University Hospital of Amiens
Locations (1):
- Activity Centre "Pain", Amiens, France

REFERENCES:
- [Result] Douleur analg. (2023) 36:73-82 DOI 10.3166/dea-2022-0249, Efficacité de la relaxation dans la fibromyalgie : un essai clinique bref aléatoirement contrôlé en simple insu portant sur 80 patients